CLINICAL TRIAL: NCT00401427
Title: A Single-centre Phase 2 Study of Vinorelbine Plus 3-weekly Trastuzumab in Metastatic Breast Cancer Overexpressing Her-2
Brief Title: HERVIN: Trastuzumab and Vinorelbine in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HERVIN
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2 overexpression; combination therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Vinorelbine

INTERVENTIONS:
Drug: trastuzumab
Drug: vinorelbine

SUMMARY:
The combination of vinorelbine with weekly trastuzumab has produced high response rate in HER2 overexpressing metastatic breast cancer (MBC). The present phase 2 study was planned to test activity of the same combination, with trastuzumab given every 3 weeks, rather than weekly.

DETAILED DESCRIPTION:
The schedule of treatment includes vinorelbine (30 mg/m2 on days 1 & 8 every 21 days) and trastuzumab (8 mg/kg on day 1 and then 6 mg/kg every 21 days). Vinorelbine is planned for maximum 9 cycles, while trastuzumab can be continued until progression. This study is a single-stage phase 2 design, and patients eligible for response evaluation are required.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer
* Stage IV
* No prior or not more than one prior chemotherapy for metastatic disease
* Overexpression of HER-2 (3+ on immunohistochemical exam) or amplified genetic expression of c-erbB2/neu (positive by Fish method)
* Performance status 0-2 (ECOG)

Exclusion Criteria:

* Absence of measurable disease
* Life expectancy < 3 months
* Concomitant malignancy or malignancy within previous 5 years (except basal cell or spinocellular skin cancer and in situ cervical cancer if they have been adequately treated
* Previous treatment with trastuzumab or vinorelbine
* Neutrophils < 1500/mm3 or platelets < 100000/mm3 or haemoglobin < 8 g/dl
* Creatinine > 1.5 x the value of the upper normal limit
* GOT and/or GPT > 2.5 x the value of the upper normal limit and/or bilirubin > 1.5 x the value of the upper normal limit in the absence of liver metastases
* GOT and/or GPT > 5 x the value of the upper normal limit and/or bilirubin > 3 x the value of the upper normal limit in the presence of liver metastases
* Left ventricular ejection fraction < 50% (measured by ultrasound or MUGA angiography)
* Concomitant conditions that contraindicate the use of the drugs in the protocol
* Male gender
* Pregnancy or lactation·
* Incapacity or refusal to provide informed consent
* Inability to comply with followup

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-11; Primary Completion 2006-06 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
response rate
toxicity

SECONDARY OUTCOMES:
time to progression
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Matteis, M.D., Principal Investigator — NCI Naples, Division of Medical Oncology C; Francesco Perrone, M.D., Ph.D., Principal Investigator — NCI Naples, Clinical Trials Unit

REFERENCES:
- [Result] De Maio E, Pacilio C, Gravina A, Morabito A, Di Rella F, Labonia V, Landi G, Nuzzo F, Rossi E, Silvestro P, Botti G, Di Bonito M, Curcio MP, Formichelli F, La Vecchia F, Staiano M, Maurea N, D'Aiuto G, D'Aiuto M, Thomas R, Signoriello G, Perrone F, de Matteis A. Vinorelbine plus 3-weekly trastuzumab in metastatic breast cancer: a single-centre phase 2 trial. BMC Cancer. 2007 Mar 20;7:50. doi: 10.1186/1471-2407-7-50. PMID 17374151